CLINICAL TRIAL: NCT03925870
Title: A Phase 2 Study to Evaluate Efficacy, Safety and Tolerability of KN046 in Subjects With Advanced Unresectable or Metastatic Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: KN046 in Subjects With Late Stage Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KN046-204
Record Dates: First submitted 2019-03-27; First posted 2019-04-24 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN046 monotherapy (Experimental): Eligible subjects will be enrolled and receive KN046 monotherapy treatment until progressive disease according to RECIST 1.1, unacceptable toxicity, completion of 2 years' KN046 treatment, or withdrawal of informed consent, whichever comes first.
  Interventions: Drug: KN046

INTERVENTIONS:
Drug: KN046 — Eligible subjects will be enrolled and receive KN046 (3 mg/kg) monotherapy treatment until progressive disease according to RECIST 1.1, unacceptable toxicity, completion of 2 years' KN046 treatment, or withdrawal of informed consent, whichever comes first

SUMMARY:
This is an open-label, multi-center, single arm study to evaluate the efficacy, safety and tolerability of KN046 in subjects with advanced unresectable or metastatic esophageal squamous cell carcinoma (ESCC).

The study is composed of 3 stages. Stage 1 (Safety run-in period) will enroll approximately 6 subjects with KN046 3 mg/kg Q2W IV, for at least 4 cycles; thereafter, Scientific Monitoring Committee (SMC) will held to review the safety profiling data and decide whether proceed to stage 2 (Expansion period). Stage 2 will enroll up to 30 subjects. After completion of the enrollment from Stage 2 and all subjects have completed at least two post baseline tumor evaluation, an interim analysis will be performed for efficacy evaluation. SMC will continuously review the safety and clinical efficacy during the study and at the interim analysis and be responsible for the decision of proceeding to Stage 3 (Biomarker enrich period).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* 18 years of age or older, Male or female,
* Pathologically confirmed diagnosis of esophageal squamous cell carcinoma (ESCC)
* Had failed at front line regimen containing fluorouracil, paclitaxel and platinum. Disease progression within 6 months from previous adjuvant chemotherapy will be considered as failure of first line systemic therapy;
* Baseline measurable disease according to RECIST 1.1 from irradiated region or progressed within a previous radiation field;
* ECOG performance status of 0 or 1;
* Have provided tumor tissue from locations not previously irradiated. Tumor biopsy may be from either the primary or metastatic site of disease;
* Adequate organ function assessed within 7 days prior to first trial treatment:
* Have a life expectancy of at least 3 months;
* If female of childbearing potential, have a negative serum pregnancy test within 7 days prior to first trial treatment;
* If female of childbearing potential or a male subject with a partner with childbearing potential, be willing to use a highly effective method of contraception (with a failure rate of less than 1.0% per year) from first study treatment to 24 weeks after completion of the trial treatment;

Exclusion Criteria:

* Untreated active CNS metastasis or leptomeningeal metastasis. Subjects may be eligible provided they are treated and clinically stable for at least 4 weeks and have no evidence of new or enlarging brain metastases and also are off steroids 7 days for treating brain metastasis prior to first trial treatment;
* Is currently participating and receiving an investigational drug or has participated in a study of an investigational drug within 4 weeks prior to the first dose of trial treatment;
* Has received other anti-tumor treatment, including traditional Chinese medicine which has approved anti-tumor indication within 4 weeks prior to the first trial treatment;
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks of the first administration of trial treatment and/or if the subject has not fully recovered from the surgery within 4 weeks of the first administration of trial treatment;
* Curative radiation within 3 months of the first dose of trial treatment. Radiation to more than 30% of the bone marrow or with a wide field of radiation should not be used within 4 weeks prior to the first administration of trial treatment;
* Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement doses, equivalent to < 10 mg prednisone daily, inhaled steroids and topical use of steroids);
* Vaccination within 28 days of the first administration of trial treatment, except for administration of inactivated vaccines (e.g., inactivated influenza vaccines);
* Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Objective response (OR) | up to 2 years
  Objective response (OR) per RECIST 1.1 criteria according to investigators assessment;
Duration of response (DOR) | up to 2 years
  Duration of response (DOR) per RECIST 1.1 criteria according to investigators assessment;

SECONDARY OUTCOMES:
Clinical benefit rate | up to 2 years
  Clinical benefit rate
Progression free survival (PFS) rates | 6 months and 12 months
  Progression free survival (PFS) rates
Overall survival (OS) rates | 6 months and 12 months
  Overall survival (OS) rates

CONTACTS AND LOCATIONS:
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China